CLINICAL TRIAL: NCT01368081
Title: A 52-week, Randomised, Multi-centre, Parallel Group Study to Investigate the Safety and Efficacy of BI 10773 (10 mg or 25 mg Administered Orally Once Daily) as add-on Therapy to an Oral Antidiabetic Drug (Sulfonylurea, Biguanide, Thiazolidinedione, Alpha Glucosidase Inhibitor, DPP-IV Inhibitor, or Glinide) in Patients With Type 2 Diabetes Mellitus With Insufficient Glycaemic Control
Brief Title: Empagliflozin (BI 10773) Comprehensive add-on Study in Japanese Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.52
Record Dates: First submitted 2011-05-19; First posted 2011-06-07 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; empagliflozin

ARMS (3):
- BI 10773 low dose (Experimental): BI 10773 low dose tablet once daily
  Interventions: Drug: BI 10773; Drug: Placebo (high dose)
- BI 10773 high dose (Experimental): BI 10773 high dose tablet once daily
  Interventions: Drug: Placebo (low dose); Drug: BI 10773
- Metformin (Active Comparator): Metformin tablets 500-2250 mg a day (twice or three times per day)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin tablets 500-2250 mg a day (twice or three times per day)
  Arms: Metformin
Drug: BI 10773 — BI 10773 low dose tablet once daily
  Arms: BI 10773 low dose
Drug: Placebo (low dose) — Placebo tablets once daily
  Arms: BI 10773 high dose
Drug: BI 10773 — BI 10773 high dose tablet once daily
  Arms: BI 10773 high dose
Drug: Placebo (high dose) — Placebo tablets once daily
  Arms: BI 10773 low dose

SUMMARY:
The objective of the study is to investigate the long-term safety and efficacy of BI 10773 given for 52 weeks as add-on therapy to one oral antidiabetic drug in patients with type 2 diabetes mellitus with insufficient glycaemic control.

ELIGIBILITY:
Inclusion criteria:

* .Diagnosis of type 2 diabetes mellitus prior to informed consent
* Male and female patients, on diet and exercise regimen, who are pre-treated with one of the following oral antidiabetic drugs: sulfonylurea, glinide, biguanide, Alpha-glucosidase inhibitor (a-GI), dipeptidyl peptidase-IV (DPP-IV) inhibitor or thiazolidinedione
* glycosylated haemoglobin (HbA1c) at Visit 1: >=7.0 to =<10.0% (national glycohemoglobin standardization program)

Exclusion criteria:

* Uncontrolled hyperglycaemia with a glucose level >240 mg/dL (>13.3 mmol/L)
* Acute coronary syndrome, stroke or transient ischemic attack (TIA) within 12 weeks prior to informed consent
* Indication of liver disease, defined by serum levels of either alanine transaminase (ALT), aspartate transaminase (AST), or alkaline phosphatase (ALP) above 3 x upper limit of normal (ULN)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1162 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (87):
- Japan (87):
  - 1245.52.023 Boehringer Ingelheim Investigational Site, Adachi-ku, Tokyo
  - 1245.52.048 Boehringer Ingelheim Investigational Site, Aki-gun, Hiroshima
  - 1245.52.012 Boehringer Ingelheim Investigational Site, Annaka, Gunma
  - 1245.52.087 Boehringer Ingelheim Investigational Site, Atami, Shizuoka
  - 1245.52.008 Boehringer Ingelheim Investigational Site, Beppu, Oita
  - 1245.52.073 Boehringer Ingelheim Investigational Site, Chiyoda-ku, Tokyo
  - 1245.52.002 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1245.52.020 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1245.52.021 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1245.52.031 Boehringer Ingelheim Investigational Site, Fujisawa, Kanagawa
  - 1245.52.077 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 1245.52.086 Boehringer Ingelheim Investigational Site, Hadano, Kanagawa
  - 1245.52.037 Boehringer Ingelheim Investigational Site, Hamamatsu, Shizuoka
  - 1245.52.046 Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - 1245.52.047 Boehringer Ingelheim Investigational Site, Hiroshima, Hiroshima
  - 1245.52.051 Boehringer Ingelheim Investigational Site, Imabari, Ehime
  - 1245.52.016 Boehringer Ingelheim Investigational Site, Iruma,Saitama
  - 1245.52.033 Boehringer Ingelheim Investigational Site, Isehara, Kanagawa
  - 1245.52.011 Boehringer Ingelheim Investigational Site, Isesaki, Gunma
  - 1245.52.045 Boehringer Ingelheim Investigational Site, Izumisano,Osaka
  - 1245.52.088 Boehringer Ingelheim Investigational Site, Kamakura, Kanagawa
  - 1245.52.072 Boehringer Ingelheim Investigational Site, Kamakura,Kanagawa
  - 1245.52.034 Boehringer Ingelheim Investigational Site, Kanazawa, Ishikawa
  - 1245.52.058 Boehringer Ingelheim Investigational Site, Kanoya, Kagoshima
  - 1245.52.019 Boehringer Ingelheim Investigational Site, Kashiwa, Chiba
  - 1245.52.039 Boehringer Ingelheim Investigational Site, Kasugai, Aichi
  - 1245.52.027 Boehringer Ingelheim Investigational Site, Kawasaki, Kanagawa
  - 1245.52.018 Boehringer Ingelheim Investigational Site, Kita-adachi-gun, Saitama
  - 1245.52.022 Boehringer Ingelheim Investigational Site, Kita-ku, Tokyo
  - 1245.52.052 Boehringer Ingelheim Investigational Site, Kitakyushu, Fukuoka
  - 1245.52.076 Boehringer Ingelheim Investigational Site, Kobe, Hyogo
  - 1245.52.026 Boehringer Ingelheim Investigational Site, Kodaira, Tokyo
  - 1245.52.069 Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - 1245.52.071 Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - 1245.52.014 Boehringer Ingelheim Investigational Site, Koshigaya, Saitama
  - 1245.52.074 Boehringer Ingelheim Investigational Site, Kuki, Saitama
  - 1245.52.055 Boehringer Ingelheim Investigational Site, Kumamoto, Kumamoto
  - 1245.52.049 Boehringer Ingelheim Investigational Site, Kure, Hiroshima
  - 1245.52.040 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 1245.52.010 Boehringer Ingelheim Investigational Site, Maebashi, Gunma
  - 1245.52.080 Boehringer Ingelheim Investigational Site, Maebashi, Gunma
  - 1245.52.050 Boehringer Ingelheim Investigational Site, Matsuyama, Ehime
  - 1245.52.075 Boehringer Ingelheim Investigational Site, Meguro-ku, Tokyo
  - 1245.52.056 Boehringer Ingelheim Investigational Site, Miyazaki, Miyazaki
  - 1245.52.057 Boehringer Ingelheim Investigational Site, Miyazaki, Miyazaki
  - 1245.52.079 Boehringer Ingelheim Investigational Site, Morioka, Iwate
  - 1245.52.003 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1245.52.004 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1245.52.005 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1245.52.038 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1245.52.059 Boehringer Ingelheim Investigational Site, Naha, Okinawa
  - 1245.52.066 Boehringer Ingelheim Investigational Site, Naha, Okinawa
  - 1245.52.065 Boehringer Ingelheim Investigational Site, Nanjyo, Okinawa
  - 1245.52.007 Boehringer Ingelheim Investigational Site, Oita, Oita
  - 1245.52.053 Boehringer Ingelheim Investigational Site, Okawa, Fukuoka
  - 1245.52.068 Boehringer Ingelheim Investigational Site, Okinawa, Okinawa
  - 1245.52.042 Boehringer Ingelheim Investigational Site, Osaka,Osaka
  - 1245.52.089 Boehringer Ingelheim Investigational Site, Osaki, Miyagi
  - 1245.52.024 Boehringer Ingelheim Investigational Site, Ota-ku, Tokyo
  - 1245.52.054 Boehringer Ingelheim Investigational Site, Saga, Saga
  - 1245.52.032 Boehringer Ingelheim Investigational Site, Sagamihara, Kanagawa
  - 1245.52.085 Boehringer Ingelheim Investigational Site, Sagamihara, Kanagawa
  - 1245.52.013 Boehringer Ingelheim Investigational Site, Saitama, Saitama
  - 1245.52.015 Boehringer Ingelheim Investigational Site, Sakado, Saitama
  - 1245.52.044 Boehringer Ingelheim Investigational Site, Sakai, Osaka
  - 1245.52.035 Boehringer Ingelheim Investigational Site, Saku, Nagano
  - 1245.52.009 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1245.52.025 Boehringer Ingelheim Investigational Site, Setagaya-ku, Tokyo
  - 1245.52.063 Boehringer Ingelheim Investigational Site, Shimajiri-gun, Okinawa
  - 1245.52.064 Boehringer Ingelheim Investigational Site, Shimajiri-gun, Okinawa
  - 1245.52.001 Boehringer Ingelheim Investigational Site, Shinjuku-ku. Tokyo
  - 1245.52.036 Boehringer Ingelheim Investigational Site, Shizuoka, Shizuoka
  - 1245.52.006 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1245.52.043 Boehringer Ingelheim Investigational Site, Takatsuki, Osaka
  - 1245.52.017 Boehringer Ingelheim Investigational Site, Tokorozawa, Saitama
  - 1245.52.070 Boehringer Ingelheim Investigational Site, Tokorozawa, Saitama
  - 1245.52.061 Boehringer Ingelheim Investigational Site, Tomigusuku, Okinawa
  - 1245.52.062 Boehringer Ingelheim Investigational Site, Tomigusuku, Okinawa
  - 1245.52.041 Boehringer Ingelheim Investigational Site, Uji, Kyoto
  - 1245.52.067 Boehringer Ingelheim Investigational Site, Uruma, Okinawa
  - 1245.52.028 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa
  - 1245.52.029 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa
  - 1245.52.030 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa
  - 1245.52.081 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa
  - 1245.52.082 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa
  - 1245.52.083 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa
  - 1245.52.084 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa

REFERENCES:
- [Derived] Shiba T, Ishii S, Okamura T, Mitsuyoshi R, Pfarr E, Koiwai K. Efficacy and safety of empagliflozin in Japanese patients with type 2 diabetes mellitus: A sub-analysis by body mass index and age of pooled data from three clinical trials. Diabetes Res Clin Pract. 2017 Sep;131:169-178. doi: 10.1016/j.diabres.2017.07.004. Epub 2017 Jul 8. PMID 28753486
- [Derived] Araki E, Tanizawa Y, Tanaka Y, Taniguchi A, Koiwai K, Kim G, Salsali A, Woerle HJ, Broedl UC. Long-term treatment with empagliflozin as add-on to oral antidiabetes therapy in Japanese patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2015 Jul;17(7):665-74. doi: 10.1111/dom.12464. Epub 2015 Apr 15. PMID 25772548

RESULTS

PARTICIPANT FLOW:
Groups:
- Sulfonylurea: Empa 10mg; Sulfonylurea: Empa 25mg: One tablet of empagliflozin (empa) once daily for 52 weeks as an add-on therapy for patients with a background treatment of Sulfonylurea
- Sulfonylurea: Metformin: 250mg tablet of metformin twice daily for 52 weeks, as an open-label treatment, for patients with background treatment of Sulfonylurea
- Biguanide: Empa 10mg; Biguanide: Empa 25mg: One tablet of empagliflozin (empa) once daily for 52 weeks as an add-on therapy for patients with a background treatment of Biguanide
- Thiazolidinedione: Empa 10mg; Thiazolidinedione: Empa 25mg: One tablet of empagliflozin (empa) once daily for 52 weeks as an add-on therapy for patients with a background treatment of Thiazolidinedione
- Alpha Glucosidase Inhibitor: Empa 10mg; Alpha Glucosidase Inhibitor: Empa 25mg: One tablet of empagliflozin (empa) once daily for 52 weeks as an add-on therapy for patients with a background treatment of Alpha glucosidase inhibitor
- DPP-IV Inhibitor: Empa 10mg; DPP-IV Inhibitor: Empa 25mg: One tablet of empagliflozin (empa) once daily for 52 weeks as an add-on therapy for patients with a background treatment of dipeptidyl peptidase IV (DPP-IV) inhibitor
- Glinide: Empa 10mg; Glinide: Empa 25mg: One tablet of empagliflozin (empa) once daily for 52 weeks as an add-on therapy for patients with a background treatment of Glinide
Period: Overall Study
Arm/Group | Sulfonylurea: Empa 10mg | Sulfonylurea: Empa 25mg | Sulfonylurea: Metformin | Biguanide: Empa 10mg | Biguanide: Empa 25mg | Thiazolidinedione: Empa 10mg | Thiazolidinedione: Empa 25mg | Alpha Glucosidase Inhibitor: Empa 10mg | Alpha Glucosidase Inhibitor: Empa 25mg | DPP-IV Inhibitor: Empa 10mg | DPP-IV Inhibitor: Empa 25mg | Glinide: Empa 10mg | Glinide: Empa 25mg
Started | 136 | 137 | 63 | 68 | 65 | 137 | 136 | 69 | 70 | 68 | 71 | 70 | 70
Completed | 126 | 128 | 59 | 63 | 63 | 127 | 124 | 62 | 62 | 58 | 62 | 67 | 63
Not Completed | 10 | 9 | 4 | 5 | 2 | 10 | 12 | 7 | 8 | 10 | 9 | 3 | 7
Not completed — Adverse Event | 4 | 4 | 3 | 2 | 2 | 5 | 6 | 2 | 3 | 5 | 6 | 1 | 3
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 4 | 1 | 1 | 0 | 3 | 4 | 2 | 5 | 4 | 3 | 2 | 0
Not completed — Other reason not defined above | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- DPP-IV Inhibitor: Empa 10mg; DPP-IV Inhibitor: Empa 25mg: One tablet of empagliflozin (empa) once daily for 52 weeks as an add-on therapy for patients with a background treatment of DPP-IV inhibitor
- Total: Total of all reporting groups
Arm/Group | Sulfonylurea: Empa 10mg | Sulfonylurea: Empa 25mg | Sulfonylurea: Metformin | Biguanide: Empa 10mg | Biguanide: Empa 25mg | Thiazolidinedione: Empa 10mg | Thiazolidinedione: Empa 25mg | Alpha Glucosidase Inhibitor: Empa 10mg | Alpha Glucosidase Inhibitor: Empa 25mg | DPP-IV Inhibitor: Empa 10mg | DPP-IV Inhibitor: Empa 25mg | Glinide: Empa 10mg | Glinide: Empa 25mg | Total
Number analyzed (Participants) | 136 | 137 | 63 | 68 | 65 | 137 | 136 | 69 | 70 | 68 | 71 | 70 | 70 | 1160
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.9) | 61.8 (9.6) | 60.0 (10.2) | 56.9 (9.5) | 57.3 (11.4) | 60.4 (10.1) | 59.7 (9.9) | 63.5 (8.8) | 61.9 (11.7) | 63.3 (9.9) | 59.1 (10.3) | 59.2 (12.1) | 57.7 (11.8) | 60.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 41 | 16 | 30 | 22 | 23 | 34 | 18 | 18 | 27 | 23 | 23 | 13 | 325
  Male | 99 | 96 | 47 | 38 | 43 | 114 | 102 | 51 | 52 | 41 | 48 | 47 | 57 | 835

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in HbA1c
Description: Change from baseline in HbA1c after 52 weeks of treatment
Time Frame: Baseline and 52 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Sulfonylurea: Empa 10mg | Sulfonylurea: Empa 25mg | Sulfonylurea: Metformin | Biguanide: Empa 10mg | Biguanide: Empa 25mg | Thiazolidinedione: Empa 10mg | Thiazolidinedione: Empa 25mg | Alpha Glucosidase Inhibitor: Empa 10mg | Alpha Glucosidase Inhibitor: Empa 25mg | DPP-IV Inhibitor: Empa 10mg | DPP-IV Inhibitor: Empa 25mg | Glinide: Empa 10mg | Glinide: Empa 25mg
Number analyzed (Participants) | 136 | 137 | 63 | 68 | 65 | 137 | 136 | 69 | 70 | 68 | 71 | 70 | 70
percentage of HbA1c | -0.93 (0.05) | -0.96 (0.05) | -0.97 (0.08) | -0.81 (0.06) | -0.98 (0.06) | -0.90 (0.05) | -0.96 (0.05) | -0.87 (0.06) | -0.77 (0.06) | -1.00 (0.06) | -0.83 (0.06) | -0.98 (0.08) | -0.98 (0.08)

2. Primary Outcome: Number of Patients With Drug Related Adverse Events
Description: Number of Patients With Drug Related Adverse Events after the first drug intake until 7 days after the last treatment administration, up to 383 days
Time Frame: After the first drug intake until 7 days after the last treatment administration, up to 383 days
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Sulfonylurea: Empa 10mg | Sulfonylurea: Empa 25mg | Sulfonylurea: Metformin | Biguanide: Empa 10mg | Biguanide: Empa 25mg | Thiazolidinedione: Empa 10mg | Thiazolidinedione: Empa 25mg | Alpha Glucosidase Inhibitor: Empa 10mg | Alpha Glucosidase Inhibitor: Empa 25mg | DPP-IV Inhibitor: Empa 10mg | DPP-IV Inhibitor: Empa 25mg | Glinide: Empa 10mg | Glinide: Empa 25mg
Number analyzed (Participants) | 136 | 137 | 63 | 68 | 65 | 137 | 136 | 69 | 70 | 68 | 71 | 70 | 70
participants | 19 | 25 | 13 | 13 | 9 | 20 | 19 | 7 | 5 | 9 | 18 | 9 | 9

3. Other Pre Specified Outcome: Confirmed Hypoglycaemic Adverse Events
Description: Number of patients with confirmed hypoglycaemic adverse events
Time Frame: After the first drug intake until 7 days after the last treatment administration, up to 383 days
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Sulfonylurea: Empa 10mg | Sulfonylurea: Empa 25mg | Sulfonylurea: Metformin | Biguanide: Empa 10mg | Biguanide: Empa 25mg | Thiazolidinedione: Empa 10mg | Thiazolidinedione: Empa 25mg | Alpha Glucosidase Inhibitor: Empa 10mg | Alpha Glucosidase Inhibitor: Empa 25mg | DPP-IV Inhibitor: Empa 10mg | DPP-IV Inhibitor: Empa 25mg | Glinide: Empa 10mg | Glinide: Empa 25mg
Number analyzed (Participants) | 136 | 137 | 63 | 68 | 65 | 137 | 136 | 69 | 70 | 68 | 71 | 70 | 70
participants | 6 | 9 | 5 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: After the first drug intake until 7 days after the last treatment administration, up to 383 days
Groups:
- Biguanide: Empa 10mg; Biguanide: Empa 25mg: tablet of empagliflozin (empa) once daily for 52 weeks as an add-on therapy for patients with a background treatment of Biguanide
- Thiazolidinedione: Empa 10mg; Thiazolidinedione: Empa 25mg: tablet of empagliflozin (empa) once daily for 52 weeks as an add-on therapy for patients with a background treatment of Thiazolidinedione
- Alpha-GI: Empa 10mg; Alpha-GI: Empa 25mg: tablet of empagliflozin (empa) once daily for 52 weeks as an add-on therapy for patients with a background treatment of Alpha-GI
- DPP-4 Inhibitor: Empa 10mg; DPP-4 Inhibitor: Empa 25mg: tablet of empagliflozin (empa) once daily for 52 weeks as an add-on therapy for patients with a background treatment of DPP-4 inhibitor
- Glinide: Empa 10mg; Glinide: Empa 25mg: tablet of empagliflozin (empa) once daily for 52 weeks as an add-on therapy for patients with a background treatment of Glinide
Arm/Group | Sulfonylurea: Empa 10mg | Sulfonylurea: Empa 25mg | Sulfonylurea: Metformin | Biguanide: Empa 10mg | Biguanide: Empa 25mg | Thiazolidinedione: Empa 10mg | Thiazolidinedione: Empa 25mg | Alpha-GI: Empa 10mg | Alpha-GI: Empa 25mg | DPP-4 Inhibitor: Empa 10mg | DPP-4 Inhibitor: Empa 25mg | Glinide: Empa 10mg | Glinide: Empa 25mg
Serious Adverse Events (participants affected / at risk) | 10/136 | 7/137 | 3/63 | 7/68 | 2/65 | 12/137 | 12/136 | 2/69 | 5/70 | 7/68 | 5/71 | 1/70 | 4/70
Other Adverse Events (participants affected / at risk) | 73/136 | 74/137 | 44/63 | 32/68 | 35/65 | 77/137 | 74/136 | 40/69 | 34/70 | 37/68 | 36/71 | 30/70 | 38/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sulfonylurea: Empa 10mg (N=136) | Sulfonylurea: Empa 25mg (N=137) | Sulfonylurea: Metformin (N=63) | Biguanide: Empa 10mg (N=68) | Biguanide: Empa 25mg (N=65) | Thiazolidinedione: Empa 10mg (N=137) | Thiazolidinedione: Empa 25mg (N=136) | Alpha-GI: Empa 10mg (N=69) | Alpha-GI: Empa 25mg (N=70) | DPP-4 Inhibitor: Empa 10mg (N=68) | DPP-4 Inhibitor: Empa 25mg (N=71) | Glinide: Empa 10mg (N=70) | Glinide: Empa 25mg (N=70)
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism arterial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Artery dissection (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukoplakia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sulfonylurea: Empa 10mg (N=136) | Sulfonylurea: Empa 25mg (N=137) | Sulfonylurea: Metformin (N=63) | Biguanide: Empa 10mg (N=68) | Biguanide: Empa 25mg (N=65) | Thiazolidinedione: Empa 10mg (N=137) | Thiazolidinedione: Empa 25mg (N=136) | Alpha-GI: Empa 10mg (N=69) | Alpha-GI: Empa 25mg (N=70) | DPP-4 Inhibitor: Empa 10mg (N=68) | DPP-4 Inhibitor: Empa 25mg (N=71) | Glinide: Empa 10mg (N=70) | Glinide: Empa 25mg (N=70)
Nasopharyngitis (Infections and infestations) | 41 | 38 | 26 | 12 | 23 | 44 | 37 | 26 | 21 | 23 | 15 | 16 | 17
Influenza (Infections and infestations) | 1 | 2 | 5 | 3 | 2 | 1 | 3 | 2 | 2 | 2 | 0 | 0 | 3
Pharyngitis (Infections and infestations) | 3 | 7 | 2 | 1 | 1 | 6 | 6 | 0 | 2 | 2 | 5 | 2 | 5
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 4 | 1 | 2 | 1 | 2 | 3 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 4 | 2 | 0 | 2 | 4 | 1 | 1 | 4 | 1 | 1 | 1 | 2
Bronchitis (Infections and infestations) | 7 | 0 | 0 | 3 | 3 | 2 | 5 | 1 | 0 | 2 | 3 | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 12 | 6 | 2 | 3 | 4 | 2 | 0 | 0 | 0 | 3 | 0 | 3
Dizziness (Nervous system disorders) | 2 | 2 | 2 | 4 | 0 | 4 | 4 | 3 | 1 | 3 | 2 | 6 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 4 | 0 | 3 | 3 | 1 | 1 | 2 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 5 | 5 | 2 | 4 | 3 | 9 | 1 | 1 | 8 | 5 | 7 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 5 | 6 | 4 | 5 | 2 | 2 | 4 | 0 | 1 | 1 | 1
Gastritis (Gastrointestinal disorders) | 3 | 2 | 2 | 1 | 1 | 4 | 2 | 2 | 4 | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 1 | 0 | 5 | 8 | 8 | 2 | 1 | 1 | 5 | 4 | 3
Pollakiuria (Renal and urinary disorders) | 3 | 6 | 0 | 2 | 0 | 11 | 3 | 2 | 3 | 4 | 7 | 3 | 5
Thirst (General disorders) | 2 | 0 | 0 | 4 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 6 | 5 | 2 | 1 | 9 | 8 | 3 | 2 | 4 | 4 | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 3 | 4 | 0 | 1 | 2 | 5 | 2 | 4 | 2 | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.